CLINICAL TRIAL: NCT05958238
Title: The Effects of Augmented Reality (AR) and Virtual Reality (VR) Oral Care Training System on Oral Healthcare for Elderly in Eldercare Students
Brief Title: The Effects of AR and VR Oral Care Training System on Oral Healthcare for Elderly in Eldercare Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-SV(I)-20230006
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Elderly; Medical Education; Augmented Reality; Virtual Reality; Oral Hygiene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AR/VR group (Experimental): Students in EG recieved a 2-hour AR/VR training for elderly oral healthcare at 2-week and 4-week follow-ups.
  Interventions: Device: AR/VR oral care training system
- Traditional teaching group (Active Comparator): Students in the CG received thirty minutes oral care training class with same teaching content in AR/VR-based training system by well-trained oral hygienist.
  Interventions: Other: Traditional classroom teaching

INTERVENTIONS:
Device: AR/VR oral care training system — Students simulated the treatment of the elderly with different physical and oral conditions using virtual situations and employed suitable oral care methods depending on each situation through VR. They learned the Bass brushing technique, the interdental brush cleaning method, and the soft tissue cleaning method through AR.
  Arms: AR/VR group
Other: Traditional classroom teaching — The well-trained oral hygienist provided traditional oral care instruction with the same teaching content in the AR/VR-based training system.
  Arms: Traditional teaching group

SUMMARY:
The aim of this study is to assess the effectiveness of an AR/VR oral care training system on the knowledge, attitudes, self-efficacy, and behavioral intentions of students majoring in geriatric care.

DETAILED DESCRIPTION:
A randomized controlled trial design will be employed, students randomly assigned to either the experimental group or the control group. The experimental group will receive a total of two sessions of AR/VR oral care training, each lasting two hours, with the intervention taking place two weeks and four weeks after completing the pre-test questionnaire. The control group, on the other hand, will receive traditional oral care instruction for thirty minutes.

Each student collected the data by a self-administered questionnaire before and immediately after each intervention.

Linear regression in generalized estimating equations (GEE) compares the differences between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Students majoring in geriatric care
* Fooyin University of Technology

Exclusion Criteria:

* Transfer student

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Oral care-related knowledge | Change from Baseline at 2-week after intervention
  20 statements were used to measure students' knowledge of the oral care of elderly. Ex: Dentures should be cleaned with toothpaste every day. With possible scores of 0-20, a higher score indicated a higher degree of oral care-related knowledge.
Oral care-related knowledge | Change from Baseline at 4-week after intervention
  20 statements were used to measure students' knowledge of the oral care of elderly. Ex: Dentures should be cleaned with toothpaste every day. With possible scores of 0-20, a higher score indicated a higher degree of oral care-related knowledge.
Attitude toward oral care | Change from Baseline at 2-week after intervention
  7 statements were used to measure students' attitude toward oral care of elderly. Ex: Oral care is as important as physical care for the elderly with disabilities. With possible scores of 7-35, a higher score indicated a more positive attitude toward oral care for elderly.
Attitude toward oral care | Change from Baseline at 4-week after intervention
  7 statements were used to measure students' attitude toward oral care of elderly. Ex: Oral care is as important as physical care for the elderly with disabilities. With possible scores of 7-35, a higher score indicated a more positive attitude toward oral care for elderly.
Self-efficacy of oral care | Change from Baseline at 2-week after intervention
  11 statements were used to evaluate students' self-efficacy in provideng the elderly with oral care. Ex: I am confident about assisting the elderly with disabilities in performing soft tissue cleaning. With possible scores of 11-55, a higher score indicated a greater degree of confidence.
Self-efficacy of oral care | Change from Baseline at 4-week after intervention
  11 statements were used to evaluate students' self-efficacy in provideng the elderly with oral care. Ex: I am confident about assisting the elderly with disabilities in performing soft tissue cleaning. With possible scores of 11-55, a higher score indicated a greater degree of confidence.
Intention to oral care behaviors | Change from Baseline at 2-week after intervention
  12 statements were used to measure students' intention to assist elderly. Ex: I will take the initiative to check the suitability of oral care tools for the elderly with disabilities. With possible scores of 12-60, a higher score indicated a higher possibility of performing the behaviors.
Intention to oral care behaviors | Change from Baseline at 4-week after intervention
  12 statements were used to measure students' intention to assist elderly. Ex: I will take the initiative to check the suitability of oral care tools for the elderly with disabilities. With possible scores of 12-60, a higher score indicated a higher possibility of performing the behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: HSIAO- LING HUANG, Dr.PH, Principal Investigator — Kaohsiung Medical University, College of Dental Medicine, Department of Oral Hygiene
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan